CLINICAL TRIAL: NCT02346344
Title: Outpatient Characterization of the Variability of Insulin Secretory Parameters in the Meal Tolerance and the Maximal Stimulation Tests of Subjects With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Foundation for the National Institutes of Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other); Amylin Pharmaceuticals, LLC. (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Eli Lilly and Company (Industry); Takeda (Industry); Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: Beta Cell - Protocol 1e
Record Dates: First submitted 2014-04-07; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; beta cell function; meal tolerance test; maximum stimulation test; method standardization; insulin secretion; prediabetes; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A multi-year clinical study to improve tools for measuring the function of insulin-producing beta cells in people with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A three-year observational study to standardize the meal tolerance and maximum stimulational tests for measuring beta cell function in the clinical setting. It also aims to improve methods for the early prediction of the long-term response to an intervention and for identification of patients at risk for rapid beta cell function deterioration, thereby enabling future clinical studies that examine diabetes progression.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent and comply with all study requirements
2. Overweight and obese men and women. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history (with the exception of glucose, see below), full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
3. T2D diagnosis by ADA criteria 2011
4. Glucose Parameters:

   1. Fasting glucose 126-270 mg/dL
   2. HbA1c 6.5%--10.0%
5. Diabetes medications allowed: metformin only: stable dose (8 weeks or longer) and 500-2000 mg/day;
6. Estimated creatinine clearance, by Cockcroft-Gault, >60 cc/min
7. No washout of medications allowed
8. Women of child-bearing potential are allowed (but must agree to use non-hormonal contraception and not plan to become pregnant for the duration of the study). Must agree to maintain the same contraceptive measures throughout the study. Acceptable contraceptive methods for female subjects of childbearing potential include one of the following:

   * Abstinence.
   * One (1) of the following methods:

     * Tubal ligation
     * Copper-containing intrauterine device (IUD)
     * Condom AND spermicidal foam/gel/film/cream/suppository
     * Male partner who has had a vasectomy for at least 6 months.
9. It is required that all male subjects use an acceptable method of contraception (as outlined below), starting from the screening period and continuing for at least 28 days after the end of the study:

   1. Abstinence
   2. A condom AND one of the following:

      * Vasectomy for more than 6 months.
      * Female partner who meets one of the following conditions:

        * Has had a tubal ligation, hysterectomy, or bilateral oophorectomy; or
        * Is post menopausal (menopause is defined as over the age of 60 years, or between 45 and 60 years being amenorrheic for at least 2 years with plasma (FSH) level > 30 UI/L) or
        * Or for female partners of the male participants, in addition to hysterectomy, oophorectorectomy, or post-menopausal status, that the use of a spermicidal gel or foam will constitute adequate protection in conjunction with use of a condom by the male.
10. BMI 27-40; stable weight (less than 3% change in past 3 months)
11. Age Range: 30-65
12. Other conditions may be allowed, if medically stable and controlled for at least four weeks within clinically acceptable limits, including: hypertension, dyslipidemia, osteoarthritis, osteoporosis
13. Smokers allowed, but must be able to participate on inpatient stay and not smoke

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, neoplastic, or allergic or clinical findings at Screening (seasonal allergies allowed).
2. Any condition possibly affecting absorption (eg, gastrectomy, malabsorption syndromes, abdominal surgery other than appendectomy, cholecystectomy or hysterectomy).
3. Use of unacceptable medications (see Appendix A)
4. A positive urine drug screen.
5. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
6. Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication.
7. 12 lead ECG demonstrating QTc >450 msec at Screening for males, 470 msec for females. If QTc exceeds 450/470 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility. An ECG with evidence for possible old myocardial infarction will need to have prior ECGs to document stability of finding.
8. Supine blood pressure >=140 mm Hg (systolic) or 90 mm Hg (diastolic), on a single measurement. If elevated, confirm by a single repeat, following at least 10 minutes of rest.
9. Screening serum alanine transaminase (ALT) or serum aspartate transaminase (AST) greater than 2X the upper limit of the laboratory reference range.
10. Elevated fasting triglycerides at screening (>500 mg/dL), confirmed by a single repeat if deemed necessary.
11. Pregnant or nursing females; inability to use effective contraception.
12. Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
13. Participation in a clinical biomedical research study within prior two months may be excluded, depending on study type and details.
14. History of sensitivity to heparin or heparin-induced thrombocytopenia, if utilized by the site for blood draws.
15. Unwilling or unable to comply with directions and procedures described in this protocol.
16. Subject is the Investigator or a sub-Investigator, research assistant, pharmacist, study coordinator, other staff, or a relative of study personnel directly involved with the conduct of the study.
17. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese individuals with type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Repeatability of the meal tolerance test and the arginine stimulation test, as indicated by the ICC (intraclass correlation coefficient) | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ruff, MD, Principal Investigator — ICON Development Solutions
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - ICON Development Solutions, Gault Lane, San Antonio, Texas